CLINICAL TRIAL: NCT05095376
Title: A Phase III Trial of Lomustine-Temozolomide Combination Therapy Versus Standard Temozolomide in Patients With Methylated MGMT Promoter Glioblastoma
Brief Title: Testing the Addition of the Chemotherapy Drug Lomustine (Gleostine) to the Usual Treatment (Temozolomide and Radiation Therapy) for Newly Diagnosed MGMT Methylated Glioblastoma
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Other - Other
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BN011; NCI-2021-10331 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN011 (Other: NRG Oncology); NRG-BN011 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Lomustine; Magnetic Resonance Spectroscopy; Photons; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (radiation therapy, temozolomide) (Active Comparator): Patients undergo radiation therapy 5 days per week and receive temozolomide PO QD for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive temozolomide PO QD on days 1-5 of each cycle. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the trial.
  Interventions: Procedure: Magnetic Resonance Imaging; Radiation: Photon Beam Radiation Therapy; Other: Questionnaire Administration; Drug: Temozolomide
- ARM II (radiation therapy, temozolomide, lomustine) (Experimental): Patients undergo radiation therapy 5 days per week for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive lomustine PO on day 1 of each cycle and temozolomide PO QD on days 2-6 of each cycle. Treatment repeats every 42 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the trial.
  Interventions: Drug: Lomustine; Procedure: Magnetic Resonance Imaging; Radiation: Photon Beam Radiation Therapy; Other: Questionnaire Administration; Drug: Temozolomide

INTERVENTIONS:
Drug: Lomustine — Given PO
  Other Names: 1-(2-Chloroethyl)-3-cyclohexyl-1-nitrosourea; 1-Nitrosourea, 1-(2-chloroethyl)-3-cyclohexyl-; Belustin; Belustine; CCNU; Cecenu; CeeNU; Chloroethylcyclohexylnitrosourea; Citostal; Gleostine; Lomeblastin; Lomustinum; Lucostin; Lucostine; N-(2-Chloroethyl)-N'-cyclohexyl-N-nitrosourea; Prava; RB-1509; WR-139017
  Arms: ARM II (radiation therapy, temozolomide, lomustine)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Photon Beam Radiation Therapy — Undergo radiation therapy
  Other Names: External beam radiation therapy using photons (procedure); Photon; Photon EBRT; Photon External Beam Radiotherapy; PHOTON Therapy; Radiation, Photon Beam
Other: Questionnaire Administration — Ancillary studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase III trial compares the effect of adding lomustine to standard chemotherapy with temozolomide and radiation therapy versus temozolomide and radiation therapy alone in shrinking or stabilizing newly diagnosed MGMT methylated glioblastoma. MGMT methylated tumors are more likely to respond to temozolomide chemotherapy. Temozolomide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill tumor cells and slow down or stop tumor growth. Lomustine is a chemotherapy drug and in a class of medications called alkylating agents. It damages the cell's DNA and may kill tumor cells. Radiation therapy uses high energy x-ray photons to kill tumor cells and shrink tumors. Adding lomustine to standard chemotherapy with temozolomide and radiation therapy may shrink or stabilize glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the regimen with the two alkylating agents temozolomide and lomustine with radiotherapy (RT) significantly prolongs overall survival (OS) versus (vs.) standard chemoradiotherapy with temozolomide in patients with newly diagnosed glioblastoma (GBM) with MGMT promoter methylation.

SECONDARY OBJECTIVES:

I. To determine if the regimen with the two alkylating agents temozolomide and lomustine with radiotherapy (RT) significantly prolongs progression-free survival (PFS) vs. standard chemoradiotherapy with temozolomide in patients with newly diagnosed GBM with MGMT promoter methylation.

II. To compare the two different chemotherapy regimens on patient-reported outcomes (PROs), as measured by the MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT) in patients with newly diagnosed GBM with MGMT promoter methylation.

III. To determine if the regimen with the two alkylating agents temozolomide and lomustine with radiotherapy (RT) is associated with inferior short-term change in PROs as measured by MDASI-BT vs. standard chemoradiotherapy with temozolomide in patients with newly diagnosed GBM with MGMT promoter methylation.

IV. To assess toxicity in the two different chemotherapy regimens.

EXPLORATORY OBJECTIVES:

I. To assess the association between absolute lymphocyte counts and outcomes. II. To assess the association between CD4+ lymphocyte counts and outcomes. III. To compare the two different chemotherapy regimens in terms of long-term PROs as measured by MDASI-BT at years 1 and 2.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo radiation therapy 5 days per week and receive temozolomide orally (PO) once daily (QD) for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive temozolomide PO QD on days 1-5 of each cycle. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo magnetic resonance imaging (MRI) throughout the trial.

ARM II: Patients undergo radiation therapy 5 days per week for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive lomustine PO on day 1 of each cycle and temozolomide PO QD on days 2-6 of each cycle. Treatment repeats every 42 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the trial.

After completion of study treatment, patients are followed up every 3 months for year 1, every 4 months for year 2, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION: No known IDH mutation. (If tested before step 1 registration, patients known to have IDH mutation in the tumor on local or other testing are ineligible and should not be registered)
* STEP 1 REGISTRATION: Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block and hematoxylin and eosin (H&E) stained slide to be sent for central pathology review for confirmation of histology and MGMT promoter methylation status. Note that tissue for central pathology review and central MGMT assessment must be received by the New York University (NYU) Center for Biospecimen Research and Development (CBRD) on or before postoperative calendar day 30. If tissue cannot be received by postoperative calendar day 30, then patients may NOT enroll on this trial as central pathology review will not be complete in time for the patient to start treatment no later than 8 weeks following surgery. Results of central pathology review and central MGMT analysis will generally be completed within 10 business days of receipt of tissue. Results will be entered by the central lab directly into Rave. Note: In the event of an additional tumor resection(s), tissue must be received within 30 days of the most recent resection and the latest resection must have been performed within 30 days after the initial resection. Surgical resection is required; stereotactic biopsy alone is not allowed because it will not provide sufficient tissue for MGMT analysis
* STEP 1 REGISTRATION: Willing to use highly effective method of contraception for participants of childbearing potential (participants who may become pregnant or who may impregnate a partner) during therapy and for 6 months after completing treatment; this inclusion is necessary because the treatment in this study may be significantly teratogenic
* STEP 1 REGISTRATION: The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information
* STEP 2 REGISTRATION: Histopathologically proven diagnosis of glioblastoma (or gliosarcoma as a subtype of glioblastoma) confirmed by central pathology review
* STEP 2 REGISTRATION: MGMT promoter with methylation confirmed by central pathology review. Note: Patients with tissue that is insufficient or inadequate for analysis, fails MGMT testing, or has indeterminate or unmethylated MGMT promoter are excluded

  * Note: Any MGMT result other than methylated would require step 2 registration to be reported as a "central review failure"
* STEP 2 REGISTRATION: Contrast-enhanced brain MRI performed either after surgery or prior to step 2 registration
* STEP 2 REGISTRATION: IDH mutation testing by at least one method (such as immunohistochemistry for IDH1 R132H) must be performed as part of standard of care and no mutation must be found (i.e IDH wildtype). (If a mutation is identified then the patient will be ineligible and must be registered as ineligible at step 2.)
* STEP 2 REGISTRATION: History/physical examination within 28 days prior to step 2 registration
* STEP 2 REGISTRATION: Karnofsky performance status (KPS) >= 70 within 28 days prior to step 2 registration
* STEP 2 REGISTRATION: Neurologic function assessment within 28 days prior to step 2 registration
* STEP 2 REGISTRATION: Age 18-70 years
* STEP 2 REGISTRATION: Hemoglobin >= 10 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 10.0 g/dl is acceptable) (Within 14 days prior to step 2 registration)
* STEP 2 REGISTRATION: Leukocytes >= 2,000/mm^3 (Within 14 days prior to step 2 registration)
* STEP 2 REGISTRATION: Absolute neutrophil count >= 1,500/mm^3 (Within 14 days prior to step 2 registration)
* STEP 2 REGISTRATION: Platelets >= 100,000/mm^3 (Within 14 days prior to step 2 registration)
* STEP 2 REGISTRATION: Total bilirubin =< 1.5 x institutional/lab upper limit of normal (ULN) (Within 14 days prior to step 2 registration)
* STEP 2 REGISTRATION: Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 2.5 x ULN (Within 14 days prior to step 2 registration)
* STEP 2 REGISTRATION: Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (Within 14 days prior to step 2 registration)
* STEP 2 REGISTRATION: Serum creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula) (Within 14 days prior to step 2 registration)
* STEP 2 REGISTRATION: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated

  * Note: Known positive test for hepatitis B virus surface antigen (HBV sAg) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy. Patients who are immune to hepatitis B (anti-hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B)
* STEP 2 REGISTRATION: For patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

  * Note: Known positive test for hepatitis C virus ribonucleic acid (HCV ribonucleic acid [RNA]) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy
* STEP 2 REGISTRATION: Known human immunodeficiency virus (HIV) infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to step 2 registration are eligible for this trial. Testing is not required for entry into protocol
* STEP 2 REGISTRATION: Negative serum or urine pregnancy test (in persons of childbearing potential) within 14 days prior to step 2 registration

  * Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal

Exclusion Criteria:

* STEP 2 REGISTRATION: Prior therapy for tumor except for resection or prior laser interstitial thermal therapy (LITT). For example, prior chemotherapy, immunotherapy, or targeted therapy for GBM or lower grade glioma is disallowed (including but not limited to temozolomide, lomustine, bevacizumab, any viral therapy, ipilimumab or other CTLA-4 antibody, PD-1 antibody, CD-137 agonist, CD40 antibody, PDL-1 or 2 antibody, vaccine therapy, polio or similar viral injection as treatment for the tumor, and/or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) as is Gliadel wafer, radiotherapy, radiosurgery, vaccine or other immunotherapy, brachytherapy, or convection enhanced delivery

  * Note: 5-aminolevulinic acid (ALA)-mediated fluorescent guided resection (FGR) photodynamic therapy (PDT) or fluorescein administered prior to/during surgery to aid resection is not exclusionary and is not considered a chemotherapy or intracerebral agent. Prior laser interstitial thermal therapy (LITT) is allowed
* STEP 2 REGISTRATION: Current or planned treatment with any other investigational agents for the study cancer
* STEP 2 REGISTRATION: Definitive clinical or radiologic evidence of metastatic disease outside the brain
* STEP 2 REGISTRATION: Prior invasive malignancy (except non-melanomatous skin cancer, cervical cancer in situ and melanoma in situ) unless disease free for a minimum of 2 years
* STEP 2 REGISTRATION: Prior radiotherapy to the head or neck that would result in overlap of radiation therapy fields
* STEP 2 REGISTRATION: Pregnancy and individuals unwilling to discontinue nursing due to the potential teratogenic effects and potential risk for adverse events in nursing infants
* STEP 2 REGISTRATION: History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide or lomustine
* STEP 2 REGISTRATION: History of pulmonary fibrosis
* STEP 2 REGISTRATION: Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring intravenous (IV) antibiotics, IV antiviral, or IV antifungal treatment
  * Symptomatic congestive heart failure, defined as New York Heart Association Functional Classification III/IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification)
  * Unstable angina pectoris within 6 months prior to Step 2 registration
  * Uncontrolled cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* STEP 2 REGISTRATION: Evidence of diffuse leptomeningeal disease that requires whole brain irradiation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-08-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From randomization to death due to any cause, assessed up to 5 years from randomization
  The Kaplan-Meier method will be used to estimate survival distribution for each treatment arm.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From randomization to disease progression or death due to any cause, whichever occurs first, assessed up to 5 years from randomization
  Analysis will consist of estimation of the PFS distribution of each treatment arm via the Kaplan-Meier method and a stratified log-rank test. Additional analyses may consist of estimating the hazard ratio via the Cox proportional hazards model, accounting for other prognostic covariates (and evaluating whether the proportional hazards assumption holds or whether any treatment effect is notably time-varying), and evaluating for potential treatment by prognostic covariate interactions.
Incidence of adverse events | Up to 5 years from randomization
  Adverse events (AEs) will be graded according to Common Terminology Criteria for Adverse Events version 5.0. Comprehensive summaries of all AEs by treatment arm will be generated and examined.
Patient reported outcomes | Up to 5 years from randomization
  Measured by the MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT) in patients with newly diagnosed glioblastoma with MGMT promoter methylation. Short-term" and "long-term" MDASI-BT, will be evaluated separately.

OTHER OUTCOMES:
Absolute lymphocyte counts | Up to 5 years from randomization
  Will assess the association between absolute lymphocyte counts and outcomes.
CD4+ lymphocyte counts | Up to 5 years from randomization
  Will assess the association between absolute lymphocyte counts and outcomes.
Estimation of the primary outcome treatment effect by sex | Up to 5 years from randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals (CIs) will be provided.
Estimation of the primary outcome treatment effect by race | Up to 5 years from randomization
  Estimates of treatment effect and the corresponding 95% CIs will be provided.
Estimation of the primary outcome treatment effect by ethnicity | Up to 5 years from randomization
  Estimates of treatment effect and the corresponding 95% CIs will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio M Iwamoto, Principal Investigator — NRG Oncology
Locations (421):
- United States (419):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - John Muir Medical Center-Concord, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Alton Memorial Hospital, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Capital Region Medical Center, Largo, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Avera Cancer Institute at Marshall, Marshall, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - John F Kennedy Medical Center, Edison, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Sands Cancer Center, Canandaigua, New York
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center in Greenville/UPMC Horizon, Greenville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Memorial Hermann Northeast Hospital, Humble, Texas
  - Memorial Hermann The Woodlands Hospital, The Woodlands, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Henrico Doctor's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (2):
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec